CLINICAL TRIAL: NCT03692455
Title: Effect of Laparoscopic Sleeve Gastrectomy Versus Roux-en-Y Gastric Bypass on Gastroesophageal Reflux Disease: An 8-Year Prospective Cohort Study.
Status: Enrolling by invitation | Type: Observational
Sponsor: Clinica Gastrobese (Other)
Collaborators: UNIVERSIDADE FEDERAL DO RIO GRANDE DO SUL (UFRGS) (Unknown)
Responsible Party: Principal Investigator, Carlos AS Madalosso, Clinical Director, Clinica Gastrobese
Other Study IDs: PP3 Folow-up
Record Dates: First submitted 2015-12-21; First posted 2018-10-02 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Gastroesophageal Reflux Disease; Morbid Obesity
Keywords: GERD; Roux-en-Y Gastric Bypass; Vertical Sleeve Gastrectomy; Lion 2.0 Consensus
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LRSYGP Group: Patients will undergo Clinical evaluation and Exams, 8 years after Laparoscopic Roux-Y Gastric Bypass.
- LSG group: Patients will undergo Clinical evaluation and Exams 8 years after Laparoscopic Sleeve Gastrectomy.

SUMMARY:
This study represents a long-term observational follow-up of patients who had previously undergone bariatric surgery (laparoscopic sleeve gastrectomy or Roux-en-Y gastric bypass) in the context of an earlier interventional trial (NCT03692455). No new interventions are assigned in the follow-up phase. Participants are evaluated clinically and functionally at predefined intervals using standardized multimodal assessments (symptom questionnaires, endoscopy, manometry, radiology, and pH monitoring).

DETAILED DESCRIPTION:
In order to determine the long term impact of Bariatric surgery on GERD, esophageal syndromes will be evaluated following the Lyon 2.0 Consensus, where troublesome symptoms were defined as score ≥ 2 on a validated questionnaire of symptoms for Portuguese language along with esophageal syndromes with injury assessed through upper endoscopy.

Esophageal acid exposure will be determined through 24h pH monitoring. Increased acid exposure will be characterized when total esophageal pH < 4 for at least 4% of its total monitoring time. The data will be collected 8 years after de surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in a previous prospective dual-cohort extension with 75 patients of the original Trial.

Original Inclusion Criteria: Inclusion criteria were age 18-70 years and body mass index (BMI) ≥40 kg/m², or ≥35 kg/m² with obesity-related comorbidities. A total of 75 patients completed the original trial.

Exclusion Criteria: Been previously submitted to any gastroesophageal surgical procedure. Presence of chronical diseases that affects esophageal motility. Do not tolerate any of the required exams

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study represents a long-term observational follow-up of 75 patients who had previously undergone bariatric surgery (laparoscopic sleeve gastrectomy or Roux-en-Y gastric bypass) in the context of an earlier interventional trial (NCT03692455). No new interventions are assigned in the follow-up phase. Participants are evaluated clinically and functionally at predefined intervals using standardized multimodal assessments (symptom questionnaires, endoscopy, manometry, radiology, and pH monitoring).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2025-10-17 (Estimated); Study Completion 2025-11-08 (Estimated)

PRIMARY OUTCOMES:
Change in number of Participants With Gastroesophageal Reflux Disease (GERD) | 8 years after intervention
  Prevalence of GERD in patients will be characterized according to Lyon 2.0 consensus

SECONDARY OUTCOMES:
Change in number of Participants Presenting GERD symptoms | 8 years after intervention
  Prevalence of typical reflux syndrome will be evaluated. In order to assess such troublesome symptoms a validated questionnaire translated into Portuguese language will be used.
Change in number of Participants With Esophageal Injury | 8 years after intervention
  Syndromes with esophageal injury should be determined exclusively by the presence of reflux esophagitis
Change in Total Esophageal Acid Exposure at 24h pH Monitoring | 8 years after intervention
  Esophageal acid exposure will be measured through 24h pH monitoring. During such period, esophageal pH will be measured and recorded as the percent of time pH stays below 4.
Change in Esophageal Acid Exposure at 24h pH Monitoring in Upright Position | 8 years after intervention
  Esophageal acid exposure will be measured through 24h pH monitoring. Esophageal pH will be measured and recorded as the percent of time pH stays below 4 while participant in upright position
Change in Esophageal Acid Exposure at 24h pH Monitoring in Supine Position | 8 years after intervention
  Esophageal acid exposure will be measured through 24h pH monitoring. Esophageal pH will be measured and recorded as the percent of time pH stays below 4 while participant in supine position
Change in number of Participants With Increased Acid Exposure | 8 years after intervention
  Increased Acid Exposure occurs when esophageal pH is <4 for a period longer than 4% of the total test time on a 24h pH monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Gursky, PhD, Study Chair — Federal University of Rio Grande do Sul
Locations (1):
- Gastrobese Clinic, Passo Fundo, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The data will be made publicly available in accordance with the requirements of the journal in which the study will be submitted